CLINICAL TRIAL: NCT00375128
Title: Assessment of Protection Against Malaria by Sporozoite Challenge of Healthy Adults Vaccinated With the Polyprotein Malaria Vaccines 'FP9-PP, MVA-PP' and Control Non-Vaccinated Volunteers
Brief Title: Sporozoite Challenge of Polyprotein Vaccinees
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Vaccine Initiative (Other)
Collaborators: University of Oxford (Other); Wellcome Trust (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC027.2; EudraCT number: 2006-000629-67; EMVI trial identifier: PP_2_04
Record Dates: First submitted 2006-09-10; First posted 2006-09-12 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Malaria, Falciparum; Malaria
Keywords: Malaria; Vaccine; Prime-boost; Challenge
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: FP9-PP (FP9 polyprotein)
Biological: MVA-PP (Modified Virus Ankara polyprotein)

SUMMARY:
This study examines the ability of two new malaria vaccines (FP9-PP and MVA-PP) to prevent the development of malaria infection after controlled exposure to the parasite. Volunteers for this trial will have received these vaccines in the preceding trial VAC027.1.

DETAILED DESCRIPTION:
Malaria infection kills over 2 million people each year. It is a major problem for those who live in endemic areas and for travellers. There is clearly a great need for a safe effective malaria vaccine.

The purpose of this study is to test the clinical efficacy of two candidate malaria vaccines (FP9-PP and MVA-PP). These live viral vector vaccines were administered in a 'prime boost' regime in the preceding trial VAC027.1.

Volunteers will now be exposed to 5 infective bites from mosquitoes carrying P. falciparum malaria.

This trial will:

1. Measure efficacy as the time in hours from malaria exposure to blood film positive for malaria parasites
2. Examine immunogenicity before and after malaria infection
3. Measure longer term vaccine efficacy by re-challenging any protected volunteers 6 - 12 months later

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-pregnant adults aged 18 to 50 years
* The vaccinated group will be subjects who have received the vaccine regime described for group 6 or 7 in VAC027.1
* Resident in or near Oxford, UK for the duration of the challenge study
* For females only, willingness to practice effective contraception during the challenge study.
* Agreement to refrain from blood donation during the course of the study
* Written informed consent
* Willingness to allow the investigators to access hospital and General Practitioner medical notes
* Willingness to undergo an HIV test

Exclusion Criteria:

* Any deviation from the protocol-defined normal range in biochemistry or haematology blood tests or in urine analysis
* Prior receipt of an investigational malaria vaccine (unless administered in VAC027.1)
* Use of any investigational or non-registered drug, live vaccine or medical device other than the study vaccine within 30 days preceding dosing of study vaccine, or planned use during the study period
* Administration of chronic immunosuppressive drugs or other immune modifying drugs within six months of vaccination
* History of malaria chemoprophylaxis with chloroquine within 5 months prior to the planned challenge, with Lariam within 6 weeks prior to the challenge, and Riamet within 2 weeks prior to the challenge
* Any history of malaria
* Travel to a malaria endemic country within the previous 3 months prior to the planned challenge
* Planned travel to malarious areas during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection and asplenia
* Evidence of cardiovascular disease
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of haemoglobinopathies
* History of diabetes mellitus
* Chronic or active neurological disease requiring ongoing specialist supervision
* Chronic gastrointestinal disease requiring ongoing specialist supervision
* History of > 2 hospitalisations for invasive bacterial infections (pneumonia, meningitis)
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Hepatomegaly, right upper quadrant abdominal pain or tenderness
* Evidence of serious psychiatric condition
* Any other on-going chronic illness requiring hospital specialist supervision
* Acute disease at the time of enrolment
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Pregnant or lactating female
* Female who is willing or intends to become pregnant during the study
* History of severe reactions or allergy to mosquito bites
* PI assessment of lack of willingness to participate and comply with all requirements of the protocol
* History or clinical evidence of intravenous drug abuse
* Any other finding which in the opinion of the investigator would significantly increase the risk of having an adverse outcome from participating in this protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26
Dates: Start 2006-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Efficacy (time in hours to parasitaemia)

SECONDARY OUTCOMES:
Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, MA, BM BCh, DPhil, DM, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Imperial College, University of London, London
  - Centre for Clinical Vaccinology & Tropical Medicine, University of Oxford, Oxford